CLINICAL TRIAL: NCT03022409
Title: A Clinical Trial to Investigate Biomarker Effects of Pre-Surgical Treatment With DDR Agents in Patients With Head and Neck Squamous Cell Carcinoma (HNSCC) Who Are Planned to Undergo Surgery That is Likely to be Followed by Radiotherapy and/or Chemotherapy.
Brief Title: A Study to Investigate Biomarker Effects of Pre-Surgical Treatment With DNA Damage Repair (DDR) Agents in Patients With Head and Neck Squamous Cell Carcinoma (HNSCC).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5330C00007
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Treatment naïve- or a second tumour; Head and Neck Squamous Cell Carcinoma (HNSCC); DNA Damage Repair (DDR)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ceralasertib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD6738 (Experimental): AZD6738 (160 mg) tablet twice daily continuous dosing for a minimum of 9 days and a maximum of 21 days.
  Interventions: Drug: Ceralasertib
- Olaparib (Experimental): Olaparib (300 mg) tablets administered orally twice daily continuously for a minimum of 9 days and a maximum of 21 days.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Ceralasertib — Ceralasertib is an oral agent and will be dosed at 160 mg. Ceralasertib tablets should be taken at the same time each day, approximately 12 hours apart (maximum ± 2 hour window) with one glass of water.
  Ceralasertib is a potent, selective inhibitor of the serine/threonine-specific protein kinase, ataxia telangiectasia and Rad3-related protein (ATR), with good selectivity against other phosphatidylinositol 3-kinase-related kinase (PIKK) family members.
  Other Names: AZD6738
  Arms: AZD6738
Drug: Olaparib — Olaparib is available as a green film-coated tablet containing 100 mg or 150 mg of Olaparib. Patients will be administered Olaparib orally twice daily at 300 mg bid. The Olaprib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Olaparib (AZD2281, KU-0059436) is a potent Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation (PARP) inhibitor (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anti-cancer agents.
  Other Names: AZD2281
  Arms: Olaparib

SUMMARY:
This biomarker study has been designed to assess the effects of different agents in both tumour tissue and peripheral samples to help inform the best combinations of DDR agents with immuno-oncology (IO) therapies. In the first instance 2 DDR agents will be assessed separately as monotherapy. Additional arms may be added later to evaluate other DDR agents and/or DDR and immunotherapy agents in combination or in sequence. The primary objective of the study is to investigate immune activation due to DDR inhibition by assessing tumour and blood samples of patients treated with study investigational agent(s).

DETAILED DESCRIPTION:
Patients are dosed for a minimum of nine days with drug. Surgery or biopsy can then take place at any time between Day 10 and Day 21 (depending on when it can be scheduled), but must occur with 24 hrs following three consecutive treatment days. During the treatment period, safety assessments must be completed at least weekly.

Follow-up will be completed after surgical resection or biopsy has been completed and can be part of standard post-surgery follow-up. If this follow-up visit occurs prior to 30 days after the final dose, a further visit or telephone call must be conducted to assess that any toxicity has resolved and to check for late toxicity.

ELIGIBILITY:
Pertinent Inclusion Criteria:

* Provision of informed consent
* Aged at least 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1 or 2 with no deterioration over the previous 2 weeks and an estimated life expectancy of greater than 12 weeks
* Treatment naïve HNSCC either newly diagnosed, or a second tumour at more than two years after successful treatment of the primary cancer, suitable for surgical resection that is likely to be followed by radiotherapy and/or chemotherapy after surgery. Patients who are suitable for radical chemoradiation without surgery are eligible if they are willing to undergo an on-treatment biopsy (FNA samples are not acceptable, specimens must be core or surgical biopsy).
* Females must be using adequate contraceptive measures, must not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential
* For the duration of the study and for 6 months after the last study drug administration, sexually active male patients must be willing to use barrier contraception i.e., condoms with all sexual partners
* No previous systemic cancer treatment or radiotherapy for the current malignancy
* Provision of genetics research informed consent

Pertinent Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous treatment with a DDR agent
* Participation in another clinical study with an investigational product during the last 21 days or 5 half-lives of the investigational product, whichever is longer
* Receiving, or having received during the week prior to first dose, corticosteroids at a dose > 10 mg prednisone/day or equivalent for any reason
* Known hypersensitivity or contraindication to any of the investigational agents or their excipients
* Small molecule investigational medicinal products (IMPs) within 28 days prior to first dose; biological IMP within 42 days prior to first dose
* Receiving, or received, concomitant medications, herbal supplements and/or foods that significantly modulate Cytochrome P450 3A4 (CYP3A4) inhibitors or moderate Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors, strong CYP3A inducers or moderate CYP3A inducers
* Impaired hepatic or renal function,inadequate bone marrow reserve or organ function
* Cardiac dysfunction defined as: Myocardial infarction within six months of study entry, New York Heart Association (NYHA) Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias or reduced LVEF < 55%
* Any of the following cardiac criteria: Mean resting corrected QTc interval using the Fridericia formula (QTcF) greater than 450 msec/male and greater than 470 msec/female or congenital long QT syndrome, clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiography (ECG), factors that increase the risk of QTc prolongation or risk of arrhythmic events, patients at risk of brain perfusion problems, relative hypotension (<100/60 mm Hg) or clinically relevant orthostatic hypotension (>20 mm Hg), uncontrolled hypertension
* Any other malignancy (i.e., non-HNSCC) which has been active or treated within the past three years (except cervical intra-epithelial neoplasia and non-melanoma skin cancer)
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection
* Judgement by the Investigator that the patient should not participate in the study
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of patient's start on the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Conversion of an immunologically based 25-gene signature from a prognostically unfavourable state to a prognostically favourable state. | From baseline through Day 31 (Follow up)
  To investigate prognosis-correlated immune activation due to DDR inhibition by monitoring the induction of immunologically relevant genes in tumours of patients treated with study investigational agent(s)

SECONDARY OUTCOMES:
Transition from a low tumour infiltrating leukocyte (TIL) state (poor prognosis) to a high TIL state (favourable prognosis) shown by TIL enumeration and an increase in CD8+ T-cells | From baseline through Day 31 (Follow up)
  To investigate the prevalence and localization of TILs associated with prognosis.
Transition from a low TIL infiltrative state (poor prognosis) to a high TIL infiltrative state (favourable prognosis) shown by TIL enumeration and an increase in CD3+ T-cells | From baseline through Day 31 (Follow up)
  To investigate the prevalence and localization of tumour infiltrating leukocytes (TILs) associated with prognosis.
Number of patients with adverse events (AE) / serious adverse events (SAE) | From time of signature of informed consent throughout the treatment period and including the follow-up period
  Assessment of the safety for each DDR agent in terms of the incidences of the AEs
Vital signs | From screening until Day 15 (+ 2 days)
  Assessment of the safety for each DDR agent in terms of the Vital signs
Clinical chemistry/haematology | From screening until Day 15 (+ 2 days)
  Assessment of the safety for each DDR agent in terms of the clinical chemistry / haematology assessments
Number of patients with abnormal findings in Electrocardiograms (ECG) | At screening and Day 1
  Assessment of the safety for each DDR agent in terms of the ECG changes. A 12-lead ECG will be performed in triplicate at screening and at a time convenient during the visits (single ECG only required at subsequent visits).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Umamaheshwar Duvvuri, Principal Investigator — University of Pittsburgh Medical Center (UPMC)
Locations (4):
- Research Site, Pittsburgh, Pennsylvania, United States
- Research Site, Toulouse, France
- Taiwan (2):
  - Research Site, Changhua
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home